CLINICAL TRIAL: NCT05252273
Title: Assessment of Patient-reported Symptoms and Endoscopic, Histologic, and Biomarker Outcomes in Patients With Acute Pouchitis Treated With Antibiotics
Brief Title: Assessment of Patients With Acute Pouchitis Treated With Antibiotics
Status: Suspended | Type: Observational
Why Stopped: This decision has been made after careful consideration and evaluation of trial progress and ongoing recruitment challenges.
Sponsor: Alimentiv Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: RCT01403
Record Dates: First submitted 2022-01-06; First posted 2022-02-23 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Pouchitis; Ulcerative Colitis
MeSH Terms: conditions — Pouchitis; Colitis, Ulcerative | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Biospecimen Retention: Samples Without DNA — * Blood collection for C-reactive protein, metabolomics, serology, proteomics, and RNA-Sequencing analyses.
  * Pouchoscopy with biopsies
  * Stool collection for microbiome, fecal calprotectin, and metabolomic analyses
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Open-label observational study: This study will evaluate the reliability and responsiveness of patient-reported symptoms and endoscopic and histologic items for assessing pouchitis disease activity in 43 patients undergoing standard of care (SOC) antibiotic therapy.
  Interventions: Other: Observational, No intervention

INTERVENTIONS:
Other: Observational, No intervention — Open-label observational study that will evaluate the reliability and responsiveness of patient-reported symptoms and endoscopic and histologic items for assessing pouchitis disease activity in 43 patients undergoing standard of care (SOC) antibiotic therapy.
  Other Names: Observational

SUMMARY:
The purpose of this study is to evaluate the reliability and responsiveness of symptoms, endoscopic, and histological items for assessing pouchitis disease activity in patients undergoing standard of care (SOC) antibiotic therapy for treatment of pouchitis, in order to develop a novel pouchitis disease activity index.

DETAILED DESCRIPTION:
This is a prospective, open-label observational study of patients with acute pouchitis being treated with SOC antibiotic therapy (a known effective therapy in most patients), to evaluate the reliability and responsiveness of existing pouchitis indices and component items for assessing pouchitis disease activity. A total of 43 subjects will be recruited and enrolled at clinical sites in North America and Europe. All subjects with suspected acute pouchitis will undergo pouchoscopy with biopsies and blood and stool sample collection at screening and receive 28 days of antibiotic therapy. Subjects will return to the clinic for a follow-up clinical assessment, pouchoscopy with biopsies forendoscopic and histologic assessments of disease activity, respectively, and blood and stool sample collection for inflammatory biomarker, molecular, and microbiome analyses approximately 6 weeks after starting antibiotic therapy. Subjects will collect an additional stool sample for fecal calprotectin (FC) and microbiome analyses and metabolomics at Week 4 and return the sample to the clinic in person or by mail. Subjects will rate their pouchitis symptoms in an electronic diary beginning at least 3 days before initiation of antibiotic therapy through to the Week 6 study visit. Total anticipated duration of subject participation is approximately 6 weeks after initiating antibiotic therapy.

Endoscopic and Histologic Disease Activity Assessments: Blinded expert endoscopists and histopathologists will serve as central readers for this study and score pouchoscopy videos and histologic slide images, respectively. Paired pouchoscopy videos and histologic slide images (baseline and Week 6) of adequate quality will be scored by central readers (see Outcome Measures). Each central reader will score all Week 6 pouchoscopy videos and histologic slide images twice, 2 weeks apart, for assessing reliability, and all baseline pouchoscopy videos/slide images once to be compared to scores posttreatment scores for assessing responsiveness.

Novel Pouchitis Disease Activity Index Development: A novel index will be developed using multiple linear regression with items that have moderate reliability and responsiveness. The index will be internally validated using the bootstrap method with 2000 replicates.

Primary Objective:

The primary objective of this study is to evaluate the reliability and responsiveness of patient-reported symptoms and endoscopic and histologic items for assessing pouchitis disease activity in patients undergoing standard of care (SOC) antibiotic therapy.

Secondary Objective:

A secondary objective of this study is to develop a novel index for assessing pouchitis disease activity.

Exploratory Objectives:

1. Identify biomarkers associated with (non)response to antibiotics in pouchitis;
2. Identify biomarkers associated with patient-reported symptoms, endoscopic, and histologic component scores and items, and pouchitis disease activity indices;
3. Describe the dynamics of the microbiome following introduction and withdrawal of antibiotics in pouchitis.

Additional exploratory analyses may be established during the review of the study results.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years of age
* IPAA for UC (J-pouch only) ≥ 6 months prior to screening
* Diagnosis of acute pouchitis at screening by stool frequency (an absolute value of ≥ 6 stools / day AND an increase of ≥ 3 stools / day above the post-IPAA baseline), and local endoscopy (presence of ≥ 1 erosion or ulceration of the pouch on endoscopy [not including ulceration occurring within 1 cm of the pouch staple or pouch suture line]).
* Not currently taking antibiotics for pouchitis or previous systemic antibiotic use for any reason within 4 weeks of screening. Prior to the Screening pouchoscopy. Note: Initiation of antibiotics for treatment of acute pouchitis prior to the Screening pouchoscopy will be permitted only if the participant initiates treatment within 48 hours prior to the Screening pouchoscopy; use outside of the 48-hour window will not be permitted and these patients should not be included in the study
* Current treatment with 5-aminosalicylic acid drugs, immunosuppressants, antidiarrheals, antimotility agents, and probiotics is permitted, if patient has received a stable dose for ≥ 4 weeks prior to screening. Dose of concomitant therapy must remain stable during the study period.
* Able to participate fully in all aspects of this clinical trial.
* Written informed consent must be obtained and documented

Exclusion Criteria:

* Pouch formations besides J-pouch (e.g., W-, S- and Kock pouches).
* IPAA for familial adenomatous polyposis.
* Pouchitis caused by other inflammatory etiologies (e.g., ischemia or infection).
* Antibiotic-dependent pouchitis, defined by ≥ 3 months of cumulative antibiotic use over the 12 months prior to screening.
* Isolated cuffitis, pouch-anal or pouch-ileal anastomotic stricture, perforating complications, or pelvic sepsis.
* Known Crohn's disease (CD) or suspected CD of the pouch, defined as complex perianal/pouch fistula and/or extensive length of prepouch ileitis with deep ulceration.
* Anticipated changes in therapy during study period.
* Use of oral corticosteroids. Participants must have discontinued oral corticosteroids within 1 month prior to screening.
* Current use of any advanced oral small molecule drug (e.g Janus kinase [JAK] inhibitors for the treatment of pouchitis. Participants must have discontinued oral small molecule therapy within 2 weeks prior to screening.
* Failed (i.e., inadequate response with, loss of response to, or intolerance to) 2 or more compounds or classes of advanced therapies such as biologics and/or small molecule drugs (i.e., 1 biologic and 1 JAK inhibitor, 2 biologics in the same class, or 2 biologics from different classes) for the treatment of pouchitis
* Participant who are pregnant or breastfeeding.
* Known history of allergy, intolerance, or are refractory to ciprofloxacin AND metronidazole AND any component of amoxicillin/potassium clavulanate combination.
* Unable to undergo endoscopic evaluation.
* Serious underlying disease other than acute pouchitis and UC that in the opinion of the investigator may interfere with the participant's ability to participate fully in the study.
* History of alcohol or drug abuse that in the opinion of the investigator may interfere with the participant's ability to comply with the study procedures.
* Prior enrollment in the current study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Forty-three subjects with acute pouchitis are to be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Estimated)
Dates: Start 2021-12-07 (Actual); Primary Completion 2024-02-12 (Estimated); Study Completion 2024-12-09 (Estimated)

PRIMARY OUTCOMES:
Change from Screening Clinical Global Impressions of Severity at Week 6 | Baseline and Week 6
  Site investigators will rate the severity of pouchitis symptoms using the Clinical Global Impressions of Severity (CGI-S) at baseline and Week 6 and change in pouchitis symptoms using the CGI of Change (CGI-C) scale at Week 6.
Change from Screening Patient's Global Impression of Severity at Week 6 | Duration of study, approximately 6 weeks.
  Participants will rate their symptoms using the Patient's Global Impression of Severity (PGI-S) at beginning at least 3 days prior to initiating antibiotic therapy through to Week 6. The weekly component will be completed at baseline and every 7 days following initiation of therapy. Change in symptoms using the PGI of Change (PGI-C) scale will be completed at Week 4 and Week 6.
Symptoms and Impacts Questionnaire for Pouchitis | Duration of study, approximately 6 weeks
  The Symptoms and Impacts Questionnaire for Pouchitis (SIQ-UC) is a self-administered tool that includes daily records of bowel movements, symptoms, and an assessment of ulcerative colitis impact on activities of daily living. For this study, the SIQ-UC has been adapted for use in pouchitis.
Visual Analog Scale for Pouchitis Symptoms | Duration of study, approximately 6 weeks
  Throughout the study, participants will rate their pouchitis symptoms daily on a 100-mm VAS,where 0 indicates "no pouchitis symptoms," and 100 indicates the "worst pouchitis symptoms ever".
Visual Analog Scale of Fecal Urgency | Duration of study, approximately 6 weeks
  Throughout the study, participants will rate fecal urgency on a 100-mm VAS, where 0 indicates "no sense of urgency to defecate" and 100 indicates "I was not able to make it to the toilet in time."
Visual Analog Scale of Abdominal Cramps Severity | Duration of study, approximately 6 weeks
  Throughout the study, participants will rate fecal urgency on a 100-mm VAS, where 0 indicates "no abdominal cramps" and 100 indicates " worst abdominal cramps ever."
Change from Baseline St. Mark's Fecal Incontinence Score (Vaizey Score) at Week 6 | Baseline and Week 6
  The St. Mark's Fecal Incontinence Score (Vaizey Score) will be completed at Screening and EOS (Week 6). Four items for incontinence and lifestyle impact are assessed on a 5-point frequency scale and 3 items are assessed with a binary yes/no response to provide a total score ranging from 0 to 24 points, with higher scores indicating greater fecal incontinence and impact on lifestyle
Endoscopic Disease Activity | Week 6
  Trained central endoscopy readers will score pouchitis endoscopic disease activity in the worst affected area of the pouch body.
Histologic Disease Activity | Week 6
  Trained central histopathology readers will score pouchitis histologic disease.

OTHER OUTCOMES:
Blood-based biomarkers of pouchitis disease activity | Baseline, Week 6
  Blood samples will be collected to identify biomarkers of pouchitis disease activity.
Stool- based biomarkers of pouchitis disease activity | Baseline, Week 4, and Week 6
  Stool samples will be collected to identify biomarkers of pouchitis disease activity.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (2):
  - Mount Sinai Hospital, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
- Toronto Immune and Digestive Health Institute (TIDHI)., Toronto, Ontario, Canada
- Academic Medical Center Amsterdam., Amsterdam, Netherlands